CLINICAL TRIAL: NCT04318262
Title: Burden of Staphylococcus Lugdunensis Infections in Hospitalized Patients: a Prospective, Bicentric Cohort Study
Brief Title: Burden of Staphylococcus Lugdunensis Infections in Hospitalized Patients
Acronym: INHOSTAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/416/OB
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Staphylococcus Lugdunensis Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Staphylococcus lugdunensis, Staphylococcus aureus or others coagulase negative Staphylococcus (CoNS) species
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient with Staphylococcus lugdunensis infection: All consecutive patients with S. lugdunensis infection (microbiological and clinical data)
  Interventions: Biological: Determination of the clinical and biological characteristics; Biological: Description of the antibiotic resistance profile; Biological: Molecular epidemiology of S. lugdunensis infections
- Patient with Staphylococcus aureus infection: Patients with S. aureus infection (microbiological and clinical data), matched to the hospital sector for S. lugdunensis infections
  Interventions: Biological: Determination of the clinical and biological characteristics; Biological: Description of the antibiotic resistance profile
- Patient with other coagulase negative Staphylococcus infection: Patients with CoNS infection (microbiological and clinical data),matched to the hospital sector for S. lugdunensis infections
  Interventions: Biological: Determination of the clinical and biological characteristics; Biological: Description of the antibiotic resistance profile

INTERVENTIONS:
Biological: Determination of the clinical and biological characteristics — * clinical data: types of infections (skin and soft tissues, bone and joint, bacteraemia, endocarditis…), delay between clinical signs and hospitalization, number of days of fever, number of days of hospitalization, infectious complications…
  * biological data: Haemoglobin, Leucocytes, Neutrophils, Creatinine clearance, CRP…
Biological: Description of the antibiotic resistance profile — Determination of MICs of the major anti-staphylococcal antibiotics by the Sensititre technique
Biological: Molecular epidemiology of S. lugdunensis infections — Genome sequencing (Illumina technique)
  Groups: Patient with Staphylococcus lugdunensis infection

SUMMARY:
Staphylococcus lugdunensis is a coagulase-negative Staphylococcus (CoNS) belonging to the normal human skin flora. It is responsible for a wide variety of infections, such as skin and soft tissue infections, bone and joint infections, but also bacteraemia and endocarditis. Although the implication of S. lugdunensis in infectious diseases is proven, many questions remain both in terms of clinical and molecular epidemiology.

In this context, INHOSTAL is the first prospective, bicentric study, which will comprehensively include all patients with S. lugdunensis infection (based on microbiological and clinical data) in two French university hospitals. The main objective of this study is thus to determine the incidence of S. lugdunensis infections in hospitalized patients.

Moreover, the originality of this project is to compare the characteristics of S. lugdunensis infections with those of infections caused by S. aureus and other species of CoNS. Thereby, the clinical epidemiology of these infections will be compared (i.e. types of infection, mode of acquisition, host risk factors…).

Finally, complete genome of all S. lugdunensis strains will be sequenced using Illumina technology and analyzed to describe the molecular epidemiology as well as the molecular mechanisms of antibiotic resistance (compared to antibiotic susceptibility evaluated by minimum inhibitory concentrations determined by Sensititre technique). This will enable to identify if predominant clones exist, and if some strains are spreading into the hospital.

The duration of the study period will be 18 months, to allow the inclusion of a total of 300 patients: 100 S. lugdunensis infections, as well as 100 S. aureus infections and 100 other species of CoNS infections.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized patients
* Patients with clinical criteria for infection
* Patients with at least one of the following microbiological criteria for infection caused by S. lugdunensis, S. aureus or other CoNS species:
* Pure culture in a normally sterile site excluding blood culture
* At least two blood cultures or one blood culture positive and a context of endocarditis or colonized material (catheter, pace-maker…)
* Pure or predominant positive culture (probable infection) in a superficial skin sample taken by swab
* At least two surgical positive cultures in case of osteo-articular infection
* Pure positive urine culture (≥104 CFU / mL), in association with abnormal leukocyturia (≥ 104 / mL)
* Patients (or trusted person) who have read the information note and who do not oppose to research participation
* Patient affiliated to the French Social Security system

Exclusion Criteria:

* Age <18 years
* Patient not affiliated to the French Social Security system
* Patient with a positive culture for S. lugdunensis, S. aureus or other CoNS species but who does not meet the inclusion criteria defined above
* Pulmonary infections of patients with cystic fibrosis
* Patient already included in the study for an infection caused by S. lugdunensis, S. aureus or other CoNS species
* Person deprived of their liberty by an administrative or judicial decision, person placed under the protection of justice, guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patient with Staphylococcus lugdunensis infection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Staphylococcus lugdunensis infections in hospitalized patients | 24 months
  Number of patients with S. lugdunensis infection during the study period, relative to the total number of patients hospitalized during the study period

SECONDARY OUTCOMES:
Clinical epidemiology of S. lugdunensis infections compared to that of S. aureus and other CoNS species | 24 months
  Comparative description of infections:
  * Clinical and biological characteristics
  * Frequency of community- and healthcare-associated infections
  * Antibiotic management and frequency of drainage and surgical procedures
  Identification of risk factors associated with infections caused by S. lugdunensis, S. aureus and other CoNS species: description of the demographic characteristics, clinical features, history of the disease, and comorbidities
Current pattern of antibiotic resistance of S. lugdunensis, S. aureus and other CoNS species | 24 months
  * For S. lugdunensis, S. aureus and other CoNS species: resistance rate to major anti-staphylococcal antibiotics according to the determination of MICs by the Sensititre technique
  * For S. lugdunensis: description of the molecular mechanisms of antibiotic resistance from whole genome sequencing data.
Molecular epidemiology of S. lugdunensis infections | 24 months
  Search for epidemic strains of S. lugdunensis in the Normandy region by comparative genomic analysis (high-throughput genome sequencing by Illumina technique)

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine DAHYOT, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Caen University Hospital, Caen
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No